CLINICAL TRIAL: NCT05532033
Title: Effect of High Flow Nasal Cannula vs Standard Oxygen Therapy on Diaphragmatic Function After Thoracic Surgery
Brief Title: High Flow Nasal Cannula and Diaphragmatic Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Fogagnolo, Principal investigator, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HFNCThoracic
Record Dates: First submitted 2022-08-09; First posted 2022-09-08 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Diaphragm Injury; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high flow nasal cannula (Experimental): Two hours after extubation patients will received high flow nasal cannula oxygenation therapy for 24 hours
  Interventions: Device: High flow nasal cannula
- Standard oxygen therapy (Active Comparator): Two hours after extubation patients will received standard oxygenation therapy for 24 hours
  Interventions: Device: Facial mask

INTERVENTIONS:
Device: High flow nasal cannula — A device able to delivery high flow oxygen therapy
  Arms: high flow nasal cannula
Device: Facial mask — standard oxygen therapy
  Arms: Standard oxygen therapy

SUMMARY:
Prospective randomized study investigating the effect of postoperative oxygen delivery on diaphragmatic function. Two different modalities of oxygen delivery will be compared: high flow nasal cannula versus standard oxygen therapy with facial mask

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective thoracic surgery

Exclusion Criteria:

* ASA score >3
* Body mass index > 35 kg/m2
* History of neuromuscular disease
* History of thoracic surgery
* Phrenic nerve paisy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
Incidence of diaphragmatic dysfunction | 24 hours after surgery
  Ultrasound evaluation of diaphragmatic dysfunction

SECONDARY OUTCOMES:
Postoperative pulmonary complication | 7 days after surgery
  Incidence of postoperative pulmonary complication

OTHER OUTCOMES:
Days without oxygen support | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study dataset will be shared in anonymous form under reasonable request
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Fogagnolo A, Grasso S, Dres M, Azzolina D, Dalla Corte F, Dolci G, Tamburini N, De Paoli G, Murgolo F, Pedarzani E, Andalo A, Volta CA, Savino S. Impact of early high flow nasal oxygen on diaphragmatic function and pulmonary complications after thoracic surgery: A randomized clinical trial. J Clin Anesth. 2025 Sep;106:111945. doi: 10.1016/j.jclinane.2025.111945. Epub 2025 Jul 23. PMID 40706477